CLINICAL TRIAL: NCT06766266
Title: A Phase I, Open-Label Clinical Study of Irinotecan Liposomes Combined with Epirubicin in Recurrent Non-Muscle Invasive Bladder Urothelium Carcinoma After Anthracyclines Treatment
Brief Title: Irinotecan Liposomes Combined with Epirubicin in Recurrent Non-muscle Invasive Bladder Urothelium Carcinoma After Anthracyclines Treatment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xin Gou, Professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-549-02
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Non-Muscle Invasive Bladder Urothelial Carcinoma

STUDY DESIGN:
Intervention Model Description: It is a double cohort study, the two cohorts are incomparable. If the recurrent tumor can't be excised by transurethral resection of bladder tumor (TURBT), the participant will enter the A arm, and if the recurrent tumor can be excised by TURBT, the participant will enter the B arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: TURBT unresectable (Experimental): If the recurrent tumor can't be excised by TURBT, participants will be assigned to this arm. Participants in this arm will complete the neoadjuvant therapy with irinotecan liposome (intravenous injection, once every two weeks for 1 month, dose increasing regimen: 37.6 mg/m2 and 56.5mg/m2) and epirubicin (intravesical instillation, once a week for 1 month, 50 mg), and the therapeutic effect was evaluated by pelvic enhanced MRI and cystoscopy. Judged by two urologists with senior professional title, patients with complete response and partial response were treated with TURBT and intravesical therapy. Patients with stable disease or progressive disease received subsequent therapy at the investigator's discretion. Participants will visit the clinic once every 2 weeks for checkups and tests.
  Interventions: Drug: Irinotecan liposome II combination therapy regimen
- Arm B: TURBT resectable (Experimental): If the recurrent tumor can be excised by TURBT, participants will be assigned to this arm (Arm B). Participants in this arm will complete TURBT with immediate intravesical instillation of epirubicin (50 mg) within 24 hours after surgery. During the induction phase (the first 1 month after surgery), participants will receive the combined therapy with irinotecan liposome (intravenous injection, once every two weeks for 1 month, dose increasing regimen: 37.6 mg/m2 and 56.5mg/m2) and epirubicin (intravesical instillation, once a week for 1 month, 50 mg). In the next 6 months, participants will continue the intravesical instillation treatment with epirubicin (once a month, 50 mg). Participants will visit the clinic once every 2 weeks for checkups and tests in the first month, and once every 3 months after the first month.
  Interventions: Drug: Irinotecan liposome II combination therapy regimen

INTERVENTIONS:
Drug: Irinotecan liposome II combination therapy regimen — In the A arm, the combined treatment with irinotecan liposome (intravenous injection, once every two weeks for 1 month, dose increasing regimen: 37.6 mg/m2 and 56.5mg/m2) and epirubicin (intravesical instillation, once a week for 1 month, 50 mg) is in the neoadjuvant therapy phase before TURBT surgery.
  Arms: Arm A: TURBT unresectable
Drug: Irinotecan liposome II combination therapy regimen — In the B arm, the combined therapy with irinotecan liposome (intravenous injection, once every two weeks for 1 month, dose increasing regimen: 37.6 mg/m2 and 56.5mg/m2 ) and epirubicin (intravesical instillation, once a week for 1 month, 50 mg) is in the induction phase after TURBT surgery.
  Arms: Arm B: TURBT resectable

SUMMARY:
The goal of this clinical trial is to learn the dose-limiting toxicity of the new combined treatment with irinotecan liposomes (intravenous injection) and epirubicin (intravesical instillation) in anthracyclines treatment-failed non-muscle invasive bladder cancer adults.

It will also learn if the combined treatment works to treat these patients. Additionally, the safety and biological mechanisms of the combined treatment will also be explored.

The main questions it aims to answer are:

* Does the combined treatment of irinotecan liposomes and epirubicin reverse anthracyclines resistance of participants?
* What medical problems do participants have after taking the combined treatment of irinotecan liposomes and epirubicin?
* What biological mechanisms underlie the effect of irinotecan liposomes on anthracyclines resistance? Participants will be classified into Arm A and Arm B.
* Arm A: Participants will receive an intravenous injection of irinotecan liposomes once every two weeks for one month, along with intravesical instillation of epirubicin once a week for one month. Patients will be evaluated by two professional urologists; those with a complete response or partial response will undergo transurethral resection of bladder tumor (TURBT) and intravesical therapy. Patients with stable or progressive disease will receive subsequent treatment at the investigator's discretion. Participants are required to visit the hospital for physical examination every two weeks.
* Arm B: In the first month after TURBT surgery, participants will receive intravenous injection of irinotecan liposomes once every two weeks for one month, and intravesical instillation of epirubicin once a week for one month, followed by once a month for six months. Participants are required to visit the clinic for physical examination once every two weeks in the first month, and once every three months after that.
* Keep a diary of their symptoms during the study period.

ELIGIBILITY:
Inclusion Criteria:

* cTa-cT1N0M0 patients with non-muscle invasive urothelial carcinoma
* Tumor recurrence occurred after anthracyclines treatment
* Systemic chemotherapy had not been used
* Tumor is measurable according to New response evaluation criteria in solid tumours: Revised RECIST guideline
* ECOG (ZPS, 5-point scale) 0-1

Exclusion Criteria:

* Age less than 18 years
* Patients with severe cardiac, cerebral, hepatic, or renal disease
* Severely malnourished patients
* Patients with mental illness and those without insight and unable to express exactly
* Combined with malignant tumors of other organs
* Systemic infectious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-04-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Bone marrow suppression (Grade four) | 4 weeks
  1. Absolute Neutrophil Count < 0.5*10^9/L
  2. Platelet <25*10^9/L
  3. leukocyte <1.0*10^9/L

SECONDARY OUTCOMES:
Safety and adverse events | 2 months
  The description of adverse events will be coded according to MedDRA terminology and graded according to NCI-CTCAE v5.0.
Objective remission rate (Arm A available) | 4 weeks
  The proportion of patients with complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) after treatment was calculated according to the recognized response evaluation criteria (such as New response evaluation criteria in solid tumours: Revised RECIST guideline , version 1.1).
  CR: All tumor target lesions disappeared and no new lesions appeared. PR: The sum of maximum diameter of tumor target lesions decreased by ≥30%; SD: The sum of the maximum diameter of tumor target lesions did not shrink to PR, or increase to PD; PD: The sum of the maximum diameters of tumor target lesions increases at least ≥20%, or new lesions appear.
Recurrence-free survival (Arm B available) | 3-6 months
  The time from TURBT surgery to recurrence or the end of follow-up.
BLM Lactylation of tumor tissues | 4 weeks
  The BLM lactylation of tumor tissue
The levels of DNA double-strand break and homologous recombination repair in tumor tissues | 4 weeks
  The levels of DNA double-strand break and homologous recombination repair in tumor tissues are detected

CONTACTS AND LOCATIONS:
Overall Officials: Xin Gou, Professor, Study Chair — cymnk@163.com
Locations (1):
- The First Affiliated Hospital of Chongqing Medica University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Yes
The study outcomes and follow-up information will be available after paper publication.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD and supporting information will be available after 2026.6.1
Access Criteria: Study protocal of the study is available from professor XinGou(email:cymnk@163.com)